CLINICAL TRIAL: NCT03328806
Title: Cross Culture Adaptation and Validation of the Arabic Version of the Core Outcome Measure Index in Patients With Low Back Pain
Brief Title: Cross Culture Adaptation and Validation of the Arabic Version of COMI in Patients With Low Back Pain
Status: Completed | Type: Observational
Sponsor: Aliaa Rehan Youssef (Other)
Responsible Party: Sponsor-Investigator, Aliaa Rehan Youssef, Assistant professor at The Department of Musculoskeletal Disorder and Its Surgery, Cairo University
Organization: Cairo University (Other)
Other Study IDs: Ay7au712017
Record Dates: First submitted 2017-09-24; First posted 2017-11-01 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Low Back Pain
Keywords: low back pain; outcome measures; cross culture adaptation; Core Outcome Measure Index
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims at translating, cross culturally adapting and establishing the psychometric properties of the The Core Outcome Measure Index (COMI) for patients with low back pain (LBP) in Egypt. This study will be conducted at the outpatient clinic of public hospitals in Egypt.

This study will be divided into two main stages: (1) Translation and cross culture adaptation, and (2) Validation.

In the translation and cross culture adaptation stage, the original English version will be translated into modern Arabic following the guidelines described by Beaton et al. (2000). Then, the translated final version will be tested on a sample of 30-40 participants in a small pilot study to ensure linguistic clarity.

For the validation stage, 100 male and female adults with LBP will be recruited from public physiotherapy outpatient clinics. Eligible patients will be asked to complete a questionnaire booklet containing The Arabic versions of Oswestry Disability index (ODI), Ronald Morris Disability Questionnaire (RMDQ), Short-form 36 (SF-36) and the Visual analogy scale (VAS).

Further, disability and function will be assessed by Timed Up and Go test (TUG), 50 feet walking and loaded reach test.

Outcome measures will include:

1. Face validity which will be evaluated subjectively based on judgment of expert committee and patients' feedback.
2. Concurrent validity is assessed by testing correlation between the COMI and VAS, ODI, RMDQ and SF-36
3. Construct validity will be assessed by testing the correlation between the scores for each item of the COMI and its corresponding valid back specific full-length questionnaire including the ODI, RMDQ, SF-36 and VAS.

All testing procedure will be repeated after seven days for testing reliability.

DETAILED DESCRIPTION:
PROCEDURE:

(1) Translation and cross culture adaptation:

The cross-cultural adaptation process for the COMI will be done as described by (Beaton et al., 2000). This will include the following phases:

1. Initial translation that includes forward translation to translate the questionnaire from the English language to Arabic by two independent bilingual translators one of them is familiar with the concepts of the COMI and the other translator doesn't have medical background. Both translators will be arabic native speakers.
2. Synthesis of the translations by comparing the two Arabic translations and combine them into one version.
3. Back translation to translate the Arabic version to the English language by two independent native english translators. It is preferred that both translator do not have any information regarding the concept being tested nor have a medical background. The two translations will be compared and a Consensus will be developed.
4. Expert committee that at least consists of a research methodologists, a health professionals, language professionals, and the translators (forward and back translators). The committee will compare between versions of the translated and original COMI and consolidate the pre-final version. The role of the expert committee to detect and correct any conceptual errors or inconsistencies, grammatical or other errors.
5. Test of the pre-final version of the instrument in a small sample (30-40 individual) to assess its content and face validity according to patients' feedback and collect comments about wording and clarity of the translated version via semi-structured interview. The sample will fulfill the study inclusion and exclusion criteria of the proposed LBP sample that will be recruited for the validation and reliability testing. Patients will be asked to complete the pre-final Arabic version of COMI and will be asked to comment on any linguistic ambiguity. Finally, researcher will discuss received comments and a consensus will be done to adapt any necessary changes.
6. Submission of documentation to the developers or coordinating committee for appraisal of the adaptation process, IN this stage all reports will be submitted at the end of the translation process to explain details of the development of each.

(2) Validation and reliability testing:

One hundred male and female adults will be recruited from public physiotherapy outpatient clinics. This sample size has been recommended as an appropriate size for reliability and validity analyses (Terwee et al., 2007). Patients will be eligible to participate in this study based on study inclusion and exclusion criteria.

Testing procedure:

First, eligible patients will have the purpose of the study and the procedures fully explained. Then, patients will be asked to participate in the study. If they accepted, an informed consent form will be signed.

Validation:

1. Concurrent validity:

   Eligible patients will be asked to complete a questionnaire booklet containing The Arabic versions of ODI, RMDQ, SF-36 and VAS.
2. Content validity:

Disability and function will be assessed by TUG, 50 feet walking and loaded reach test (Bennell, et al., 2011). All tests will be demonstrated to the patient in details before asking them to take the test as follow:

Timed Up and Go test (TUG):

First, a 3-meter distance will be marked on the floor. An armchair will be placed at one end of this distance. This test will be performed by measuring the time (in seconds) required by the patients to stand from sitting position and walk at his/her normal pace then turn back to the starting position(Bohannon, 2006; Herman and Hausdorff, 2011).

50-feet walk test: The patient will walk 25 foot forward then return back to the starting position as fast as s/he could. The time spent in this task will be measured in seconds using a stopwatch (Simmonds et al., 1998)

ELIGIBILITY:
Inclusion Criteria:

1. Adults male and females with age ranging from 21 to 50 years.
2. Referred with a diagnosis of low back pain described as pain and discomfort, localized below the costal margin and above the inferior gluteal folds, with or without referred leg pain (Airaksinen et al., 2006).
3. Arabic speaking in the Egyptian dialect.

Exclusion Criteria:

1. Back pain secondary to known specific pathology (e.g. infection, tumor, Osteoporosis, fracture, structural deformity, inflammatory disorder (e.g. ankylosing spondylitis), radicular syndrome or cauda equine syndrome) (Mannion et al., 2012).
2. Pregnant women
3. Post-operative patients
4. Patients who had traumatic injury in the lower quadrant within the past 6 months.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will be delimited to:
  1-140 Egyptian patients diagnosed clinically with LBP with or without leg pain. 2- Patients' age ranging from 21 years to 50
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Correlation between the COMI and Ronald Morris Disability Questionnaire (RMDQ) | 1 day
  This will be done to assess the construct validity. RMDQ evaluates the disability associated with LBP. It consists of 24 yes/no items related specifically to physical functions including walking, bending over, sitting, lying down, dressing sleeping, self-care and daily activities. Patients are asked whether the statements apply to them that day (i.e. the last 24 h). One point is given for each item. The total score ranges from 0 (no disability) to 24 (severe disability).

SECONDARY OUTCOMES:
Correlation between the COMI and Visual Analogue Scale (VAS) | 1 day
  To assess concurrent validity. The VAS is a valid and reliable scale to assess pain. It ranges from 0 (no pain) to 10 (severe excruciating pain). Pain will be given a line measuring 10 com, with 0 and 10 marked on opposite ends. Then, patient will be asked to put a mark on that line to indicate the level of pain experienced.
Correlation between the COMI and Oswestry Disability Index (ODI) | 1 day
  To assess concurrent validity. ODI is a self-reported questionnaire consisting of questions arranged in 10 domains. Each domain contains six questions that are scored ranging from 0 (minimum degree of difficulty in that activity) to 5 (maximum degree of difficulty). These questions assess the activities of daily living in patients with LBP, including pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and travelling. If more than one statement is marked in each section, the highest score should be taken. The total score is 50 which expressed as a percentage.
Correlation between the COMI and Short Form 36 (SF-36) | 1 day
  To assess concurrent validity. SF-36 is a short-form questionnaire for measuring health surveys (physical, role, and social functioning, mental health, and general health perceptions) and two concepts were added by empirical work (bodily pain and vitality).
Perceived changes in back and/or leg pain | 1 day
  Patients will be asked to report any change in current back or leg pain at the time of second testing using a 5-point Likert scale (a little bit better, better, no chance, a little bit worse, worse)
Reliability of COMI | 7-14 days
  Patients will be asked to complete COMI after seven to 14 days days to test its reliability by comparing between the results at the first and second time to detect any discrepancies.
Face validity | 1 day
  The face validity is dependent on judgment of expert committee and patients' feedback.

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa Rehan Youssef, PhD, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Faculty of Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al-Disoky S, El-Ghoul Y, Heissam K, & Mohamed R. Prevalence of Low Back Pain and its Effect on Quality of Life among Patients Attending Abokhalefa Center, Ismailia Governorate. Med. J. Cairo Univ, 83(1), 385-394, 2015.
- [Background] Duthey B. Background paper 6.24 low back pain. World Health Organisation (WHO)(ed.) Priority medicines for Europe and the world 'A public health approach to innovation'. Geneva: WHO. 2013 Mar 15.
- [Background] Andresen EM. Criteria for assessing the tools of disability outcomes research. Arch Phys Med Rehabil. 2000 Dec;81(12 Suppl 2):S15-20. doi: 10.1053/apmr.2000.20619. PMID 11128900
- [Background] Nakhostin Ansari N, Naghdi S, Eskandari Z, Salsabili N, Kordi R, Hasson S. Reliability and validity of the Persian adaptation of the Core Outcome Measure Index in patients with chronic low back pain. J Orthop Sci. 2016 Nov;21(6):723-726. doi: 10.1016/j.jos.2016.07.022. Epub 2016 Aug 18. PMID 27545452
- [Background] Atlas SJ, Deyo RA. Evaluating and managing acute low back pain in the primary care setting. J Gen Intern Med. 2001 Feb;16(2):120-31. doi: 10.1111/j.1525-1497.2001.91141.x. PMID 11251764
- [Background] Azimi, P. Comparing COMI and RMDQ-24, NCOS, ODI, JOA and SSS Questionnaires in Patients with Lumbar Spinal Stenosis. WSCJ, 3: 87-90, 2012
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Bennell K, Dobson F, Hinman R. Measures of physical performance assessments: Self-Paced Walk Test (SPWT), Stair Climb Test (SCT), Six-Minute Walk Test (6MWT), Chair Stand Test (CST), Timed Up & Go (TUG), Sock Test, Lift and Carry Test (LCT), and Car Task. Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S350-70. doi: 10.1002/acr.20538. No abstract available. PMID 22588756
- [Background] Beurskens AJ, de Vet HC, Koke AJ, van der Heijden GJ, Knipschild PG. Measuring the functional status of patients with low back pain. Assessment of the quality of four disease-specific questionnaires. Spine (Phila Pa 1976). 1995 May 1;20(9):1017-28. doi: 10.1097/00007632-199505000-00008. PMID 7631231
- [Background] Bohannon RW. Reference values for the timed up and go test: a descriptive meta-analysis. J Geriatr Phys Ther. 2006;29(2):64-8. doi: 10.1519/00139143-200608000-00004. PMID 16914068
- [Background] Chou YC, Shih CC, Lin JG, Chen TL, Liao CC. Low back pain associated with sociodemographic factors, lifestyle and osteoporosis: a population-based study. J Rehabil Med. 2013 Jan;45(1):76-80. doi: 10.2340/16501977-1070. PMID 23052969
- [Background] Costa LO, Maher CG, Latimer J. Self-report outcome measures for low back pain: searching for international cross-cultural adaptations. Spine (Phila Pa 1976). 2007 Apr 20;32(9):1028-37. doi: 10.1097/01.brs.0000261024.27926.0f. PMID 17450079
- [Background] Damasceno LH, Rocha PA, Barbosa ES, Barros CA, Canto FT, Defino HL, Mannion AF. Cross-cultural adaptation and assessment of the reliability and validity of the Core Outcome Measures Index (COMI) for the Brazilian-Portuguese language. Eur Spine J. 2012 Jul;21(7):1273-82. doi: 10.1007/s00586-011-2100-3. Epub 2011 Dec 15. PMID 22170447
- [Background] Deyo RA, Battie M, Beurskens AJ, Bombardier C, Croft P, Koes B, Malmivaara A, Roland M, Von Korff M, Waddell G. Outcome measures for low back pain research. A proposal for standardized use. Spine (Phila Pa 1976). 1998 Sep 15;23(18):2003-13. doi: 10.1097/00007632-199809150-00018. PMID 9779535
- [Background] Eisenberg DM, Davis RB, Ettner SL, Appel S, Wilkey S, Van Rompay M, Kessler RC. Trends in alternative medicine use in the United States, 1990-1997: results of a follow-up national survey. JAMA. 1998 Nov 11;280(18):1569-75. doi: 10.1001/jama.280.18.1569. PMID 9820257
- [Background] Elders LA, Burdorf A. Prevalence, incidence, and recurrence of low back pain in scaffolders during a 3-year follow-up study. Spine (Phila Pa 1976). 2004 Mar 15;29(6):E101-6. doi: 10.1097/01.brs.0000115125.60331.72. PMID 15014283
- [Background] Ferrer M, Pellise F, Escudero O, Alvarez L, Pont A, Alonso J, Deyo R. Validation of a minimum outcome core set in the evaluation of patients with back pain. Spine (Phila Pa 1976). 2006 May 20;31(12):1372-9; discussion 1380. doi: 10.1097/01.brs.0000218477.53318.bc. PMID 16721302
- [Background] Genevay S, Cedraschi C, Marty M, Rozenberg S, De Goumoens P, Faundez A, Balague F, Porchet F, Mannion AF. Reliability and validity of the cross-culturally adapted French version of the Core Outcome Measures Index (COMI) in patients with low back pain. Eur Spine J. 2012 Jan;21(1):130-7. doi: 10.1007/s00586-011-1992-2. Epub 2011 Sep 1. PMID 21881865
- [Background] Grotle M, Brox JI, Vollestad NK. Functional status and disability questionnaires: what do they assess? A systematic review of back-specific outcome questionnaires. Spine (Phila Pa 1976). 2005 Jan 1;30(1):130-40. PMID 15626993
- [Background] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034
- [Background] Hall AM, Maher CG, Latimer J, Ferreira ML, Costa LO. The patient-specific functional scale is more responsive than the Roland Morris disability questionnaire when activity limitation is low. Eur Spine J. 2011 Jan;20(1):79-86. doi: 10.1007/s00586-010-1521-8. Epub 2010 Jul 14. PMID 20628767
- [Background] Heneweer H, Vanhees L, Picavet HS. Physical activity and low back pain: a U-shaped relation? Pain. 2009 May;143(1-2):21-5. doi: 10.1016/j.pain.2008.12.033. Epub 2009 Feb 12. PMID 19217208
- [Background] Herman T, Giladi N, Hausdorff JM. Properties of the 'timed up and go' test: more than meets the eye. Gerontology. 2011;57(3):203-10. doi: 10.1159/000314963. Epub 2010 May 20. PMID 20484884
- [Background] Kaila-Kangas L, Keskimaki I, Notkola V, Mutanen P, Riihimaki H, Leino-Arjas P. How consistently distributed are the socioeconomic differences in severe back morbidity by age and gender? A population based study of hospitalisation among Finnish employees. Occup Environ Med. 2006 Apr;63(4):278-82. doi: 10.1136/oem.2005.021642. PMID 16556749
- [Background] Kessler JT, Melloh M, Zweig T, Aghayev E, Roder C. Development of a documentation instrument for the conservative treatment of spinal disorders in the International Spine Registry, Spine Tango. Eur Spine J. 2011 Mar;20(3):369-79. doi: 10.1007/s00586-010-1474-y. Epub 2010 Jun 9. PMID 20532924
- [Background] Lee CE, Simmonds MJ, Novy DM, Jones S. Self-reports and clinician-measured physical function among patients with low back pain: a comparison. Arch Phys Med Rehabil. 2001 Feb;82(2):227-31. doi: 10.1053/apmr.2001.18214. PMID 11239315
- [Background] Lozano-Alvarez C, Perez-Prieto D, Salo G, Molina A, Llado A, Ramirez M. Usefulness of the core outcome measures index in daily clinical practice for assessing patients with degenerative lumbar disease. Adv Orthop. 2012;2012:474685. doi: 10.1155/2012/474685. Epub 2012 Mar 5. PMID 22518325
- [Background] Mannion AF, Balague F, Pellise F, Cedraschi C. Pain measurement in patients with low back pain. Nat Clin Pract Rheumatol. 2007 Nov;3(11):610-8. doi: 10.1038/ncprheum0646. PMID 17968331
- [Background] Mannion AF, Boneschi M, Teli M, Luca A, Zaina F, Negrini S, Schulz PJ. Reliability and validity of the cross-culturally adapted Italian version of the Core Outcome Measures Index. Eur Spine J. 2012 Aug;21 Suppl 6(Suppl 6):S737-49. doi: 10.1007/s00586-011-1741-6. Epub 2011 Mar 17. PMID 21409562
- [Background] Mannion AF, Elfering A, Staerkle R, Junge A, Grob D, Semmer NK, Jacobshagen N, Dvorak J, Boos N. Outcome assessment in low back pain: how low can you go? Eur Spine J. 2005 Dec;14(10):1014-26. doi: 10.1007/s00586-005-0911-9. Epub 2005 Jun 4. PMID 15937673
- [Background] Mannion AF, Porchet F, Kleinstuck FS, Lattig F, Jeszenszky D, Bartanusz V, Dvorak J, Grob D. The quality of spine surgery from the patient's perspective. Part 1: the Core Outcome Measures Index in clinical practice. Eur Spine J. 2009 Aug;18 Suppl 3(Suppl 3):367-73. doi: 10.1007/s00586-009-0942-8. Epub 2009 Mar 25. PMID 19319578
- [Background] Mannion AF, Vila-Casademunt A, Domingo-Sabat M, Wunderlin S, Pellise F, Bago J, Acaroglu E, Alanay A, Perez-Grueso FS, Obeid I, Kleinstuck FS; European Spine Study Group (ESSG). The Core Outcome Measures Index (COMI) is a responsive instrument for assessing the outcome of treatment for adult spinal deformity. Eur Spine J. 2016 Aug;25(8):2638-48. doi: 10.1007/s00586-015-4292-4. Epub 2015 Oct 30. PMID 26519374
- [Background] McHorney CA, Ware JE Jr, Raczek AE. The MOS 36-Item Short-Form Health Survey (SF-36): II. Psychometric and clinical tests of validity in measuring physical and mental health constructs. Med Care. 1993 Mar;31(3):247-63. doi: 10.1097/00005650-199303000-00006. PMID 8450681
- [Background] Mehlum IS, Kristensen P, Kjuus H, Wergeland E. Are occupational factors important determinants of socioeconomic inequalities in musculoskeletal pain? Scand J Work Environ Health. 2008 Aug;34(4):250-9. doi: 10.5271/sjweh.1269. Epub 2008 Sep 22. PMID 18815713
- [Background] Miekisiak G, Banach M, Kiwic G, Kubaszewski L, Kaczmarczyk J, Sulewski A, Kloc W, Libionka W, Latka D, Kollataj M, Zaluski R. Reliability and validity of the Polish version of the Core Outcome Measures Index for the neck. Eur Spine J. 2014 Apr;23(4):898-903. doi: 10.1007/s00586-013-3129-2. Epub 2013 Dec 23. PMID 24363040
- [Background] Nicholas MK. The pain self-efficacy questionnaire: Taking pain into account. Eur J Pain. 2007 Feb;11(2):153-63. doi: 10.1016/j.ejpain.2005.12.008. Epub 2006 Jan 30. PMID 16446108
- [Background] Qiao J, Zhu F, Zhu Z, Xu L, Wang B, Yu Y, Qian BP, Ding Y, Qiu Y. Validation of the Simplified Chinese version of the Core Outcome Measures Index (COMI). Eur Spine J. 2013 Dec;22(12):2821-6. doi: 10.1007/s00586-013-2761-1. Epub 2013 Apr 3. PMID 23549908
- [Background] Rubin DI. Epidemiology and risk factors for spine pain. Neurol Clin. 2007 May;25(2):353-71. doi: 10.1016/j.ncl.2007.01.004. PMID 17445733
- [Background] Simmonds MJ, Olson SL, Jones S, Hussein T, Lee CE, Novy D, Radwan H. Psychometric characteristics and clinical usefulness of physical performance tests in patients with low back pain. Spine (Phila Pa 1976). 1998 Nov 15;23(22):2412-21. doi: 10.1097/00007632-199811150-00011. PMID 9836355
- [Background] Smeets R, Koke A, Lin CW, Ferreira M, Demoulin C. Measures of function in low back pain/disorders: Low Back Pain Rating Scale (LBPRS), Oswestry Disability Index (ODI), Progressive Isoinertial Lifting Evaluation (PILE), Quebec Back Pain Disability Scale (QBPDS), and Roland-Morris Disability Questionnaire (RDQ). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S158-73. doi: 10.1002/acr.20542. No abstract available. PMID 22588742
- [Background] Soliman T. Activities of daily living as a parameter of pain relief in low back patient. Master Thesis, Alexandria University, Faculty of Medicine, 1999.
- [Background] Storheim K, Brox JI, Lochting I, Werner EL, Grotle M. Cross-cultural adaptation and validation of the Norwegian version of the Core Outcome Measures Index for low back pain. Eur Spine J. 2012 Dec;21(12):2539-49. doi: 10.1007/s00586-012-2393-x. Epub 2012 Jun 14. PMID 22695701
- [Background] Terwee CB, Bot SD, de Boer MR, van der Windt DA, Knol DL, Dekker J, Bouter LM, de Vet HC. Quality criteria were proposed for measurement properties of health status questionnaires. J Clin Epidemiol. 2007 Jan;60(1):34-42. doi: 10.1016/j.jclinepi.2006.03.012. Epub 2006 Aug 24. PMID 17161752
- [Background] Thomas E, Silman AJ, Croft PR, Papageorgiou AC, Jayson MI, Macfarlane GJ. Predicting who develops chronic low back pain in primary care: a prospective study. BMJ. 1999 Jun 19;318(7199):1662-7. doi: 10.1136/bmj.318.7199.1662. PMID 10373170
- [Background] Turk DC, Dworkin RH, Allen RR, Bellamy N, Brandenburg N, Carr DB, Cleeland C, Dionne R, Farrar JT, Galer BS, Hewitt DJ, Jadad AR, Katz NP, Kramer LD, Manning DC, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robinson JP, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Witter J. Core outcome domains for chronic pain clinical trials: IMMPACT recommendations. Pain. 2003 Dec;106(3):337-345. doi: 10.1016/j.pain.2003.08.001. PMID 14659516
- [Background] Von Korff M, Simon G. The relationship between pain and depression. Br J Psychiatry Suppl. 1996 Jun;(30):101-8. PMID 8864155
- [Background] Waxman R, Tennant A, Helliwell P. A prospective follow-up study of low back pain in the community. Spine (Phila Pa 1976). 2000 Aug 15;25(16):2085-90. doi: 10.1097/00007632-200008150-00013. PMID 10954640
- [Background] Webb R, Brammah T, Lunt M, Urwin M, Allison T, Symmons D. Prevalence and predictors of intense, chronic, and disabling neck and back pain in the UK general population. Spine (Phila Pa 1976). 2003 Jun 1;28(11):1195-202. doi: 10.1097/01.BRS.0000067430.49169.01. PMID 12782992